CLINICAL TRIAL: NCT04428931
Title: Evaluation of Attentional Performance in Parkinson Disease
Brief Title: Attentional Performance in Parkinson Disease
Status: Withdrawn | Type: Observational
Why Stopped: The pandemic caused a delay in starting the study; PI is leaving.
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 200102; 20-N-0102
Record Dates: First submitted 2020-06-11; First posted 2020-06-11 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Parkinson's Disease
Keywords: Functional Connectivity; Visual Attention; Dopamine Depletion; Landmark Test
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- PD patients: Patients with Asymmetric Parkinson's disease

SUMMARY:
Background:

Parkinson Disease (PD) is a nervous system disorder that affects movement. Dopamine is an important neurotransmitter in the brain. As PD progresses, there is less and less dopamine in the brain. Researchers think there may be a relationship between differences in attention and dopamine in people with PD.

Objective:

To learn if people with PD that is worse on one side also have differences in how much attention they pay to the two sides of space on their left and right.

Eligibility:

English-speaking, right-handed people age 35-80 with PD.

Design:

Participants will be screened with medical and neurological history and exam, and medicine review.

Participants will have 1 study visit. It will last 7-8 hours. They will stop taking their Parkinson medicine 12 hours before the visit.

Participants will complete questionnaires.

Participants will do tasks on a computer screen. They will judge the middle of lines, react to stimuli, and search and identify items that appear on the screen.

Participants may have functional and structural magnetic resonance imaging (MRI). MRI uses a strong magnetic field and radio waves to take pictures of the brain. During the MRI, participants will lie on a table that slides in and out of the MRI scanner. While inside the scanner, they will look at a cross on a screen, relax, and think about nothing.

Participants will undergo prism adaptation. They will sit in front of a board while their chin rests on a support. They will point to 1 of 2 dots on the board while they wear prism glasses that shift their vision to the left or right....

DETAILED DESCRIPTION:
Study Description:

We will investigate the relationship between Dopamine (DA) function and attention in patients with asymmetric Parkinson Disease (PD). We hypothesize that the direction of asymmetry in dopamine (DA) depletion predicts the asymmetry in visual attention.

Objectives:

Primary Objective:

- to study attentional asymmetry in patients with PD. We hypothesize that visual attention in Parkinson will be biased to the visual field contralateral to the least affected hemisphere (i.e. contralateral to the most affected side).

Secondary Objectives:

* to investigate the correlation between feedback learning and visuospatial attention performance in PD. We hypothesize that feedback learning will also be affected according to the most compromised hemisphere. Right hemisphere-predominant PD patients (left-motor predominant), compared to left hemisphere-predominant patients, will exhibit a rightward visuospatial bias and a relative preference for learning from reward, compared to punishment.
* to investigate the effect of prism adaptation on feedback learning and visuospatial attention in PD. This objective is exploratory.

Endpoints:

Primary Endpoint: visuospatial performance on the Landmark Task

Secondary Endpoints: performance on:

* Posner Task
* Visual Search Task
* Attentional blink Task
* Visuospatial performance on the Manual Line Bisection Task
* Reward and Punishment Implicit Feedback Learning Task
* The Attentional Scaling Task

Functional connectivity measured with resting state fMRI.

Study Population:

Sixty patients with asymmetric PD. Any gender, aged 35-80 (inclusive), able to give consent and without a diagnosis of significant illness affecting the central nervous system other than PD.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Provision of signed and dated informed consent form
  2. Stated willingness to comply with all study procedures and availability for the duration of the study
  3. Male or female aged 35 - 80 (inclusive)
  4. Fluent in English
  5. Right-handed per the Edinburgh Handedness scale
  6. Able to provide consent
  7. Diagnosis of idiopathic Parkinson s disease according to UK Brain Bank criteria
  8. On dopaminergic therapy to treat Parkinsonian symptoms
  9. MOCA Score greater than or equal to 24 determined by a NIH neurologist
  10. Hoehn and Yahr Score less than or equal to 3 determined by a NIH neurologist
  11. Asymmetric motor symptoms

EXCLUSION CRITERIA:

1. Any current major neurological or psychiatric disorder other than Parkinson s disease, such as, (but not limited to) stroke, dementia, Alzheimer disease, Schizophrenia or Major Depression Disorder
2. Inability to provide consent
3. Members of the Behavioral Neurology Unit, NINDS
4. Left-handed per the Edinburgh Handedness scale
5. Primarily axial motor symptoms or symmetrical limb involvement
6. Pregnancy
7. Exclusion criteria for MRI

   * Presence of metal which would make having an MRI scan unsafe, such as pacemakers, stimulators, pumps, aneurysm clips, metallic prostheses, artificial heart valves, cochlear implants or shrapnel fragments, or if subject was a welder or metal worker, since small metal fragments may be present in the eye.
   * Claustrophobia
   * Inability to lie supine comfortably for 1 hour
   * Pregnancy

INCLUSION OF VULNERABLE PARTICIPANTS:

Because the goals of the study can be accomplished without involving vulnerable population, we will not include individuals without consent capacity.

Since the goal is to characterize visuospatial attention deficits in idiopathic PD which is a disease of late adulthood, we will not include children.

The effects of MRI on fetal development and the health of pregnant women is unknown.

Therefore, women who are pregnant and breast-feeding will be excluded and women who can become pregnant will be excluded following a positive pregnancy test, if the optional MRI is under consideration.

The study requires fluency in English in order to completely understand tasks instructions, thus non-English speakers/readers will be excluded.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asymmetric PD patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2021-12-06 (Actual)

PRIMARY OUTCOMES:
Attentional asymmetry | 2 months
  Direction and degree of visuospatial bias on the Landmark task

SECONDARY OUTCOMES:
Feedback learning and visuospatial attention performance | 2 months
  Direction and degree of visuospatial bias on the Manual Line Bisection, Visual Search Posner, Attentional Blink, Reward and Punishment Implicit Feedback Learning, and the Attentional Scaling Tasks

CONTACTS AND LOCATIONS:
Overall Officials: Eric M Wassermann, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-N-0102.html